CLINICAL TRIAL: NCT05581446
Title: The Effects of Pain Types on Pain Severity and Quality of Life in Chronic Neck Pain
Brief Title: Pain Types and Pain Severity in Chronic Neck Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-15/19
Record Dates: First submitted 2022-10-10; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Chronic Neck Pain
MeSH Terms: interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Visual Analogue Scale — pain type severity determination and quality of life assessment
  Other Names: Pain Catastrophizing Scale; Neck Disability İndex; short form-36; painDETECT; Clinical criteria and rating score for nociplastic pain affecting the musculoskeletal system

SUMMARY:
The aim of this study is to characterize the distribution of pain phenotypes in people with chronic neck pain and to determine the effects of pain phenotypes on pain severity, functional status and quality of life.

Participants will be examined to determine the type of pain and questions will be asked to assess pain severity and impact.

ELIGIBILITY:
Inclusion Criteria:

* having chronic neck pain
* be over 18 years old

Exclusion Criteria:

* those under the age of 18
* Those with major psychiatric illness,
* Those with communication problems

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients presenting with chronic neck pain
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
identification of pain types(determination of nociceptive, neuropathic, nociplastic pain rates) | 01.06.2023
  Neuropathic pain with PainDETECT scale, Clinical criteria and rating system for nociplastic pain affecting the musculoskeletal system nosplastic pain will be evaluated
determination of pain intensity and effects(Pain severity,quality of life,disability,pain status) | 01.06.2023
  Pain severity with Visual Analogue Scale, quality of life with SF-36, disability with Neck Disability İndex, pain status with Pain Catastrophizing Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Beyhekim Research and Training Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Will be shared if requested.

REFERENCES:
- [Derived] Akkurt HE, Karpuz S, Yilmaz R, Gures F, Gures SC, Erol K, Yilmaz H. The effects of pain types on pain intensity and quality of life according to the mechanism in chronic neck pain. Saudi Med J. 2025 Jun;46(6):695-701. doi: 10.15537/smj.2025.46.6.20240394. PMID 40516931